CLINICAL TRIAL: NCT04464512
Title: Suboxone User Perioperative Early Referral and Enhanced Recovery After Surgery- Orthopaedic Trauma Surgery Population
Acronym: SUPER-ERAS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No qualified enrollments; study cancelled due to pandemic
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Michael Kyle Ritchie, Assitant Professory of Anesthesiology, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1802003669
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Addiction Opiate; Chronic Pain; Fractures, Bone; Buprenorphine Dependence
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain; Fractures, Bone | interventions — Sufentanil; Buprenorphine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant is blind to the treatment/group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (control) treatment (No Intervention): The control group receives 1mcg/kg fentanyl followed by fentanyl 0.5-1mcg/kg q10 minute PRN, ketorolac 0.5mg/kg up to 30mg max IV, and acetaminophen 1000mg IV for pain control intraoperatively. The patient is then treated with hydromorphone 0.005mg/kg q10minutes the post-anesthesia recovery. The patient would then receive hydromorphone 0.005 mg/kg q1hr PRN, 1 gram acetaminophen IV scheduled q6hr, and methocarbamol 750mg QID following discharge from the PACU and transfer to the hospital floor. The patient is converted to oxycodone 10mg (Roxicodone) q4hr PRN and 975 mg PO APAP scheduled for pain control on postoperative day number 1 or when appropriate for PO intake. The patients receives their home dose of suboxone onpostoperative day number 1 or when appropriate for PO intake.
  On postoperative day number 2 number 3, patients are transitioned to an increased dose of their Suboxone for pain control in preparation for discharge.
- Treatment Group (Active Comparator): Buprenorphine-sufentanil group receives sufentanil 0.03mcg/kg followed by sufentanil 0.01-0.03 mcg/kg q10 min PRN, IV ketorolac 0.5mg/kg up to 30mg max and IV acetaminophen 15mg/kg up to 1000mg for pain control intraoperatively. In the PACU, IV buprenorphine 0.3mg IV q30 minutes would be given as the first line choice for pain control for 3 doses. IV PCA sufentanil is used as a second line therapy if patient comfort is not achieved by IV buprenorphine alone. The patient receives 0.3 mg buprenorphine IV Q6hr PRN, scheduled IV acetaminophen 1 gram for 24 hrs and methocarbamol 750mg QID after discharge from the PACU and transfer to the floor. The patient is converted to buprenorphine2mg q6hr PRN and 975 gram PO APAP scheduled for pain control on postoperative day 1. The patient receives their home dose of Suboxone starting on postoperative day 1 if tolerating PO intake. On postoperative day 2, patients would be transitioned to an increased dose of their Suboxone.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — IV buprenorphine plus IV sufentanil treatment group.
  Other Names: Buprenorphine
  Arms: Treatment Group

SUMMARY:
This is a randomized controlled trial. Patients will be randomly assigned to either the control or treatment group, with equal allocation using block randomization. The primary null hypothesis is that a combination sufentanil and buprenorphine based pain control regimen will not result in lower morphine equivalent requirements for pain control when compared to a classic fentanyl and hydromorphone based regimen. The secondary working hypothesis is that the patient satisfaction survey mean satisfaction scores will be higher in the buprenorphine and sufentanil treated group when compared to the classic fentanyl and hydropmorphone treated group. The secondary null hypothesis is that the patient satisfaction surveys mean scores will not be significantly different in the buprenorphine and sufentanil treated group when compared to the classic fentanyl and hydropmorphone treated group. The tertiary working hypothesis is that the patients will have significantly lower rates of relapse as defined by follow up with their home suboxone clinic at 2 and 4 weeks. The tertiary null hypothesis is that patients have equivalent rates of relapse as defined by follow up with their home suboxone clinic at 2 and 4 weeks.

DETAILED DESCRIPTION:
After determining the patient qualifies for the study, the patient would then be taken through the informed consent process by one of the co-investigators in the orthopedics group at West Virginia University. The co-investigator would then use a block randomization table to assign the patient to standard (control) treatment versus IV buprenorphine plus IV sufentanil treatment group. The appropriate order set would then be selected in EPIC by the anesthesia department depending on the results of the randomization. Induction of anesthesia, anxiolysis and hypnosis would be at the discretion of the assigned anesthesiologist. Ketamine would be excluded as an option for maintenance of general anesthesia due to its profound analgesic properties. The control group would receive fentanyl 0.5mcg/kg q10 minute PRN, ketorolac 0.5mg/kg up to 30mg max IV, and acetaminophen 1000mg IV for pain control intraoperatively. The patient would then be treated with hydromorphone 0.005mg/kg q10 minutes (max single dose 1mg) in the post-anesthesia recovery unit (PACU) until their pain was described as manageable or the patient reported they were comfortable. The patient would then receive hydromorphone 0.005 mg/kg (max single dose 1mg) q1hr PRN, 1 gram acetaminophen IV scheduled q6hr, and methocarbamol 750mg QID following discharge from the PACU and transfer to the hospital floor. The patient would then be converted to oxymorphone 10mg (Roxicodone) q4hr PRN and 975 mg PO APAP scheduled for pain control on hospital day number 2. The patients would receive their home dose of suboxone on hospital day number 2. On hospital day number 3, patients would be transitioned to an increased dose of their Suboxone for pain control in preparation for discharge. At any time during admission the patient feels as if their pain is uncontrolled and comfort could not be achieved, the anesthesia pain service would evaluate the patient and order sufentanil PCA while discontinuing other opioid therapy. This treatment would be considered a rescue therapy and the patient would be removed from the study arm. The buprenorphine-sufentanil group would receive sufentanil 0.01 mcg/kg q10 min PRN, IV ketorolac 0.5mg/kg up to 30mg max and IV acetaminophen 15mg/kg up to 1000mg for pain control intraoperatively. In the PACU, IV buprenorphine 0.3mg IV q30 minutes would be given as the first line choice for pain control for 3 doses. IV PCA sufentanil would be used as a second line therapy if patient comfort is not achieved by IV buprenorphine alone. The patient would then receive 0.3 mg buprenorphine IV Q6hr PRN, scheduled IV acetaminophen 1 gram for 24 hours and methocarbamol 750mg QID after discharge from the PACU and transfer to the hospital floor on hospital day 1. The patient would then be converted to buprenorphine 2mg q6hr PRN and 975 gram PO APAP scheduled for pain control on hospital day number 2. The patient would receive their home dose of suboxone starting on hospital day number 2. On hospital day number 3, patients would be transitioned to an increased dose of their suboxone for pain control as determined by psychiatry in preparation for discharge.

Post-operatively both groups would receive psychiatric consult and PT/OT consult. Data on opioid consumption for the intra-operative period and post-operative period as well as post-operative pain scores will be recorded and analyzed for comparison. Morphine equivalents used per hour and per 24 hours would be analyzed as a primary endpoint. A patient pain satisfaction survey would be distributed and collected from both groups on hospital day #3. Data on length of stay, pain scores, and ED readmission for pain control would also be recorded and analyzed. Patients would be discharged on increased dose suboxone for 2 weeks for post-operative pain control. The patients would then transition back to their normal suboxone maintenance dose. A follow up phone call would be made at 2 and 4 weeks to the home clinic to assess patient follow up and potential relapse.

Univariate statistics (e.g. mean, median, standard deviation, interquartile range) will be used to summarize the collected data. Balance between the two groups for key patient variables will be assessed using a two-sided two-sample t-test using unequal variances and the Welch modification to the degrees of freedom. For categorical variables, the Chi-square test will be used. If non-parametric tests or exact methods are required, the Mann-Whitney U test and the Fisher exact test will be used as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic trauma patient with history of suboxone use for greater than 30 days. Trauma must involve major long bone fracture(s) (femur, tibia, fibula, humerus, radius, ulna) .Must have taken suboxone in the last 24 hours and have participated in addiction treatment for greater than one month.
* Age 18-65
* ASA I-III
* Willing to participate in post-operative psychiatric care
* Glascow Coma Scale 15

Exclusion Criteria:

* Severe renal disease (Creatinine clearance < 40)
* History of chronicSevere liver disease or an (AST/ALT greater than 2 times normal, direct/indirect bilirubin outside normal limits and INR> 1.4 if drawn as standard of care) or evidence of acute liver failure
* Acute Ethanol Intoxication (serum ethanol > 0.080 at time of informed consent)
* Severe distracting injury that is close to pain levels expected from the orthopedic trauma (Ex surgical abdominal process, neurosurgical process, massive soft tissue trauma, severe spinal injury, multiple rib fractures)
* Pregnancy
* Polysubstance abuse on urine or serum drug screen (excluding marijuana due to its new legality in multiple states)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Pain Medication Used | up to 4 weeks
  Total amount of pain medication used

SECONDARY OUTCOMES:
Patient Satisfaction Survey Results | Post operative day number 2
  Patient will complete a satisfaction survey on day 2

CONTACTS AND LOCATIONS:
Locations (1):
- West Viriginia University Hospital, Morgantown, West Virginia, United States